CLINICAL TRIAL: NCT07004361
Title: Ethical Issues of Using Gene Therapy in the Treatment of AMD (Age-related Macular Degeneration)
Brief Title: Ethical Issues of Using Gene Therapy in the Treatment of AMD
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_HM_001
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: ethical; Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to examine the legitimacy of gene therapy use in the treatment of exudative age-related macular degeneration (AMD). This involves questioning its beneficence/non-maleficence ratio given the limited experience with this innovative technology and its irreversible effects, requiring a surgical procedure for administration. Additionally, the study explores patient autonomy in decision-making concerning complex therapeutic approaches and how patients should be supported to best uphold this autonomy.

DETAILED DESCRIPTION:
Qualitative research based on semi-structured interviews conducted with patients diagnosed with age-related macular degeneration (AMD), followed in the ophthalmology department of Nantes University Hospital and treated with intravitreal injections. These interviews are structured around three main themes in order to better understand:

The experience and perception of the current treatment by the patients

Their perceptions, expectations, and potential concerns regarding gene therapy

Their perception and understanding of decision-making autonomy in their health decisions

ELIGIBILITY:
Inclusion Criteria:

* Patients with exsudative AMD, male female >18 years Patients for whom the doctor could consider gene therapy.

Exclusion Criteria:

Patients with atrophic AMD (Age-related Macular Degeneration) Patients with other degenerative retinal diseases than AMD, Patients with with associated cognitive disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: exsudative AMD patients in o^pthalmology department in CHU Nantes
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The experience and current treatment outcomes perceived by patients | 1 months
  Semi-structured interviews

SECONDARY OUTCOMES:
Patients' perceptions, expectations, and potential concerns regarding gene therapy | 1 month
  Semi-structured interviews
Patients' perception and representation of decisional autonomy in their health decisions | 1 month
  Semi-structured interviews